CLINICAL TRIAL: NCT03700502
Title: Use Resting-state Functional Magnetic Resonance Imaging (Rs-fMRI) to Explore the Brain Activity in Patients With Painful Diabetic Neuropathy (PDN) in Order to Study Central Mechanism of PDN.
Brief Title: Functional Magnetic Resonance Imaging of Brain Activity in Patients With Painful Diabetic Neuropathy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Collaborators: Jiangsu Province Nanjing Brain Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201605027
Record Dates: First submitted 2018-09-27; First posted 2018-10-09 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-03

CONDITIONS: Painful Diabetic Neuropathy
Keywords: resting state functional MRI; painful diabetic neuropathy
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- patients with painful diabetic neuropathy
  Interventions: Diagnostic Test: resting-state functional Magnetic Resonance Imaging
- diabetics with non-pain neuropathy
  Interventions: Diagnostic Test: resting-state functional Magnetic Resonance Imaging
- gender and age matched healthy controls
  Interventions: Diagnostic Test: resting-state functional Magnetic Resonance Imaging

INTERVENTIONS:
Diagnostic Test: resting-state functional Magnetic Resonance Imaging — The investigators used fraction Amplitude of Low Frequency Fluctuation (fALFF) and Regional Homogeneity (ReHo) of resting-state functional Magnetic Resonance Imaging (rs-fMRI) to explore the brain activity in patients with PDN in order to study the central mechanism. The investigators also evaluated the symptoms, signs and mental conditions of the patients.

SUMMARY:
Patients with painful diabetic neuropathy (PDN) often combine with anxiety and depression. However, the pathogenesis of PDN is unclear, especially the mechanism associated with central nervous system. The investigators used fraction Amplitude of Low Frequency Fluctuation (fALFF) and Regional Homogeneity (ReHo) of resting-state functional Magnetic Resonance Imaging (rs-fMRI) to explore the brain activity in patients with PDN in order to study the central mechanism.The investigators evaluated the symptoms, signs and mental conditions of patients with PDN and non-pain neuropathy. The brain Blood Oxygen Level Dependent (BOLD) fMRI scan was performed in patients together with some gender and age matched healthy controls. Maybe this study can find that patients with PDN have abnormal brain activity, indicating central nervous system may contribute to painful diabetic neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation and signing informed consent
* 18 to 60 years old with junior high school education or above
* meeting the 1999 WHO type 2 diabetes diagnostic criteria: having symptoms of diabetes (polydipsia, polyphagia, polyuria and unexplained weight loss) plus one of the following 3 items: (1) random blood glucose more than 11.1 mmol/L; (2) fasting blood glucose more than 7 mmol/L; (3) after 2 hours glucose load, the blood sugar more than 11.1 mmol/L
* The diagnosis of diabetic peripheral neuropathy (at the same time meets the following three items, of which painful neuropathy patients have pain symptom): (1) neuropathy occurs not earlier than the diagnosis of diabetes; (2) having clinical manifestations of pain, numbness, and abnormal sensation; (3) any abnormality in the following 5 examinations: ankle reflex, vibratory sensation, pressure sensation, temperature sensation, and acupuncture pain

Exclusion Criteria:

* left-hand writers
* neuropathy caused by other causes, such as cervical spondylosis, cerebral infarction, Green Barre syndrome; severe arteriovenous disease; neurotoxic changes caused by drugs and renal insufficiency
* patients with severe cerebral vascular disease
* diagnosed mental disorders such as depression, anxiety and Alzheimer's disease
* patients who can't accept head magnetic resonance imaging, such as those with metal (stents, metal dentures, internal fixation plates, etc.), and claustrophobic space phobias

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Meet the diagnosis of diabetic peripheral neuropathy (at the same time meets the following three items, of which painful neuropathy patients have pain symptom): (1) neuropathy occurs not earlier than the diagnosis of diabetes; (2) having clinical manifestations of pain, numbness, and abnormal sensation; (3) any abnormality in the following 5 examinations: ankle reflex, vibratory sensation, pressure sensation, temperature sensation, and acupuncture pain.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-06-05 (Actual); Primary Completion 2018-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
resting-state functional Magnetic Resonance Imaging | one or two years
  collect and analyze the data of brain fMRI

CONTACTS AND LOCATIONS:
Locations (1):
- the first hospital of Nanjing, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Liu X, Xu X, Mao C, Zhang P, Zhang Q, Jiang L, Yang Y, Ma J, Ye L, Lee KO, Wu J, Yao Z. Increased thalamo-cortical functional connectivity in patients with diabetic painful neuropathy: A resting-state functional MRI study. Exp Ther Med. 2021 May;21(5):509. doi: 10.3892/etm.2021.9940. Epub 2021 Mar 19. PMID 33791018
- [Derived] Zhang Q, Zhang P, Yan R, Xu X, Mao C, Liu X, Li F, Ma J, Ye L, Yao Z, Wu J. A Single-Blinded Trial Using Resting-State Functional Magnetic Resonance Imaging of Brain Activity in Patients with Type 2 Diabetes and Painful Neuropathy. Diabetes Ther. 2019 Feb;10(1):135-147. doi: 10.1007/s13300-018-0534-x. Epub 2018 Nov 30. PMID 30506341